CLINICAL TRIAL: NCT06095258
Title: A Practical Clinical Randomized Controlled Trial of Traditional Chinese Medicine in the Treatment of Long COVID and an Analysis of Syndrome Types and Medication Characteristics of Traditional Chinese Medicine
Brief Title: A Practical RCT of TCM in the Treatment of LCOVID and Analysis of Syndrome Types and Medication Characteristics.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhang Hongwei, Dr., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parametric LCOVID
Record Dates: First submitted 2023-10-20; First posted 2023-10-23 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Long COVID
Keywords: Traditional Chinese medicine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Intervention Model Description: Totally 162 patients with long COVID recruited into the study will be randomly assigned to the traditional Chinese medicine treatment group or the Western medicine control group. Patients in the treatment group will receive individualized TCM syndrome differentiation treatment, and patients in the control group will receive conventional Western medicine symptomatic treatment from general Western medicine practitioners.
Who Masked: Outcomes Assessor
Masking Description: The outcome data collectors are blinded throughout the study. Patients will be specifically instructed not to disclose specific treatment received to outcome data collectors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese medicine treatment group (Experimental): Patients in this treatment group will receive individualized TCM syndrome differentiation treatment.
  Interventions: Drug: Traditional Chinese medicine treatment
- Western medicine control group (Active Comparator): Patients in this control group will receive conventional Western medicine symptomatic treatment from general Western medicine practitioners.
  Interventions: Drug: Western medicine treatment

INTERVENTIONS:
Drug: Traditional Chinese medicine treatment — About four to six Chinese medicine practitioners with five to twenty years of clinical work experience will be responsible for patient diagnosis and prescription treatment, and use a uniformly designed data collection form to record the patient's medical history, clinical symptoms and signs, tongue and pulse conditions, and other information. Patients in the treatment group will receive individualized Chinese medicine treatment prescriptions. Patients in the control group received conventional Western medicine treatment, and about 3 to four Western medicine practitioners with five to twenty years of work experience will be responsible for the conventional medicine prescription. The treatment of the two groups will last for four weeks, and the patients will be followed up for four weeks after the treatment. A patient diary will be provided to all participants for recording the drug compliance and any adverse event during the treatment period.
  Other Names: CM group
  Arms: Traditional Chinese medicine treatment group
Drug: Western medicine treatment — Western medicine doctors will mainly use symptomatic drugs to treat long COVID. For example, cough medicine (such as codeine), bronchodilators (such as ventolin), expectorants (such as fluimucil) and so on are used to treat cough, shortness of breath, or other respiratory symptoms. Non-steroidal anti-inflammatory painkillers (such as panadol) are often used for treating headaches, and sedative-hypnotic drugs (such as stilnox) are often used to treat insomnia.
  Other Names: WM group
  Arms: Western medicine control group

SUMMARY:
This is a multi-center, outcome assessor-blinded, practical randomized controlled trial, aiming to compare the actual clinical effectiveness of individualized traditional Chinese medicine and conventional Western medicine in the treatment of long COVID.

Totally 162 patients with long COVID recruited into the study will be randomly assigned to the traditional Chinese medicine treatment group or the Western medicine control group. Patients in the treatment group will receive individualized TCM syndrome differentiation treatment, and patients in the control group will receive conventional Western medicine symptomatic treatment from general Western medicine practitioners for 4 weeks. All patients were followed up once a week (±2 days) during treatment period and followed up by 4 weeks (±2 days) after the treatment. Outcome measurements will be conducted at baseline, the end of treatment (week 4 ±2 days) and the follow-up visit (week 8 ±2 days).

DETAILED DESCRIPTION:
The novel coronavirus has caused a global pandemic since the end of 2019. As of November 27, 2022, 637 million people have been diagnosed worldwide and more than 6 million people have died. Studies have reported that about 10%-20% of people will continue to have some post-infection symptoms after being infected with the new coronavirus. The World Health Organization (WHO) named it the Post COVID-19 Condition or Long COVID. The main symptoms of Long COVID include severe fatigue, shortness of breath, heart damage (such as myocarditis), cognitive impairment, sleep disturbance, post-traumatic stress disorder syndrome, muscle pain, decreased concentration, headache, impaired taste, and smell, etc.

In the face of the ongoing epidemic and more and more people being infected, people are increasingly concerned about the long-term impact of the new coronavirus infection. At present, western medicine is trying to adopt symptomatic treatment for some main symptoms of COVID-19. In addition, people are also trying many non-drug treatments, such as exercise, pulmonary rehabilitation training, cognitive behavioral therapy, etc.

Traditional Chinese medicine (TCM) has been strongly involved in the treatment and prevention of COVID-19 and the recovery of COVID-19 infection in the early stages of the epidemic. In order to cope with the fifth wave of the epidemic in Hong Kong, in April 2022, the Chinese government's Anti-epidemic Chinese Medicine Expert Group in Hong Kong launched the "Guidelines on the Rehabilitation of Traditional Chinese Medicine during the Recovery Period of Coronavirus Disease 2019 (Trial Version)". However, there is a lack of clinical research evidence that has practical guiding value for the TCM syndrome diagnosis and medication in long COVID patients. Secondly, there is a lack of reliable research evidence on the clinical effectiveness of individualized Chinese medicine treatment of long COVID. Thirdly, there is a lack of large-scale research data on patients with long COVID from clinical treatment. Fourthly, there is a lack of comparative research evidence between traditional Chinese medicine and conventional Western medicine.

Therefore, this study will be conducted in order to understand the possible advantages or disadvantages of traditional Chinese medicine compared with Western medicine; improve the efficacy of traditional Chinese medicine in the treatment of long COVID; and promote the application of traditional Chinese medicine in the field of long COVID treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects with age between 6 and 80 years old;
* For those who have recovered from COVID-19, it has been more than 28 days since the date of diagnosis (the diagnosis is confirmed by rapid antigen test or positive nucleic acid test of deep throat saliva or nose/throat swab);
* The average score of the modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) is above 2 (i.e. above the moderate level).

Exclusion Criteria:

* People who have not been infected with COVID-19;
* People who are still positive for COVID-19;
* Known history of some certain serious medical disease, which is in an unstable state or even affects basic survival, such as cardiovascular disease, liver or renal dysfunction, diabetes, cancer, cerebrovascular disease, blood disorders;
* Known impaired hematological characteristics or impaired liver/kidney function;
* People with mild cognitive impairment, that is, those whose age/education matching percentile in the score of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) is lower than 16; or those who cannot truthfully fill out the questionnaire due to mental and psychological factors;
* Have used any drugs or other treatment methods for the treatment of COVID-19 in the past week, such as acupuncture, massage, scraping, cupping, etc.;
* Known history of allergy to any traditional Chinese medicine.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
5-level EQ-5D version (EQ-5D-5L) | 4 weeks
  The 5-level EQ-5D version (EQ-5D-5L) was developed by the European Society for Quality of Life (EuroQol) and has been validated [38]. The EQ-5D-5L assesses a patient's quality of life by assessing five dimensions: mobility, self-care, daily activities, pain or discomfort, and anxiety or depression. Each aspect is assessed by 5 levels, namely none, mild, moderate, heavy, and very severe. In addition, patients self-rated their overall health status using a visual analog scale (EQVAS).
5-level EQ-5D version (EQ-5D-5L) | 8 weeks
  The 5-level EQ-5D version (EQ-5D-5L) was developed by the European Society for Quality of Life (EuroQol) and has been validated [38]. The EQ-5D-5L assesses a patient's quality of life by assessing five dimensions: mobility, self-care, daily activities, pain or discomfort, and anxiety or depression. Each aspect is assessed by 5 levels, namely none, mild, moderate, heavy, and very severe. In addition, patients self-rated their overall health status using a visual analog scale (EQVAS).

SECONDARY OUTCOMES:
Measure Yourself Medical Outcome Profile in Chinese version (CMYMOP2) | 4 weeks
  The Chinese version of the Measure Yourself Medical Outcome Profile has been validated [39]. This questionnaire asks respondents to name one or two symptoms of greatest concern and the daily activities that are limited by these symptoms. Respondents rate these symptoms and activities, as well as their general health status, on a scale from 0 to 6 (0 is best, 6 is worst).
Measure Yourself Medical Outcome Profile in Chinese version (CMYMOP2) | 8 weeks
  The Chinese version of the Measure Yourself Medical Outcome Profile has been validated [39]. This questionnaire asks respondents to name one or two symptoms of greatest concern and the daily activities that are limited by these symptoms. Respondents rate these symptoms and activities, as well as their general health status, on a scale from 0 to 6 (0 is best, 6 is worst).
Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) | 4 weeks
  This improved version of the scale allows patients to self-assess the main symptoms of the COVID, the degree of functional limitation and overall health status. There are 17 items in total, including shortness of breath, cough/throat sensitivity/voice change, fatigue, changes in smell or taste, pain or discomfort, and cognition. problems, palpitations/dizziness, tiredness/exacerbation after work, anxiety/depression, sleep problems, communication, walking or moving, self-care, other daily activities, social roles), and other symptoms (such as fever, hair loss, dry eyes, tinnitus, nausea, etc.) and general health, etc. Each item is scored from 0 to 3 (0 is asymptomatic, 1 is mild and does not affect daily life, 2 is moderate and affects daily life to a certain extent, and 3 is severe or affects daily life comprehensively).
Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) | 8 weeks
  This improved version of the scale allows patients to self-assess the main symptoms of the COVID, the degree of functional limitation and overall health status. There are 17 items in total, including shortness of breath, cough/throat sensitivity/voice change, fatigue, changes in smell or taste, pain or discomfort, and cognition. problems, palpitations/dizziness, tiredness/exacerbation after work, anxiety/depression, sleep problems, communication, walking or moving, self-care, other daily activities, social roles), and other symptoms (such as fever, hair loss, dry eyes, tinnitus, nausea, etc.) and general health, etc. Each item is scored from 0 to 3 (0 is asymptomatic, 1 is mild and does not affect daily life, 2 is moderate and affects daily life to a certain extent, and 3 is severe or affects daily life comprehensively).
Serum level change of inflammatory factors | 4 weeks
  Inflammatory markers including interferon (IFN-β), interferon (IFN-λ2/3), pentraxin 3 (PTX3) and interleukin 6 will be measured.
Safety assessment | 4 weeks
  In order to evaluate the safety of the traditional Chinese medicine treatment, the patient's complete blood count (CBC) and liver and kidney function indicators will be tested before starting the study treatment and after the treatment ends.
Adverse event | 4 weeks
  Subjects will be asked about the occurrence of any adverse events during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhang, PhD, Principal Investigator — School of Chinese Medicine